Official Title: SOVA Ambassadors Community Setting

NCT number: NCT06066697

Date of document creation: 8/23/2023

Date of last modification: 9/24/2025

STUDY TITLE
SOVA Ambassadors Community Setting

Ы

Dr. Ana Radovic

Study Coordinator Contact information

Email: <a href="mailto:sovalab@pitt.edu">sovalab@pitt.edu</a>
Phone: 412-368-2619

**FUNDING SOURCE** 

National Institute on Minority Health and Health Disparities

### STUDY INFORMATION

This is a research study using the SOVA website which is a website for youth mental health education. The research study will compare two interventions for young people ages 14 to 21 who participate in workforce development programs. We are recruiting 40 young people.

This study takes about 12 weeks. Participants will take a baseline survey, a 6-week survey, and a 12 week survey.

After you complete the first survey (or baseline), we will then randomize you into one of the two groups. Randomization by the computer is like flipping a coin to decide which group you will be in.

In <u>Group 1</u> or the SOVA Ambassador arm you will get access to the SOVA website as a content creator. You will provide a username and email you would like to use for the website. The research assistant will create a login for you for the site and give you information about what it means to participate as a SOVA Ambassador including information about compensation, expectations, and procedures. Expectations include that at least once a month for three months you will contribute an entry for the website. This entry may be an article that you write yourself (a blog post) or you can also choose to have a ghostwriter – this would mean the research assistant meets with you to interview you about a topic and then writes an article about it without using any private info about you and has you approve it first before its posted. The entry can also be a photo, video, or music (without identifying information or images) about mental health.

SOVA Ambassadors follow a set of ground rules such as not to post any identifying information on the site to keep the site anonymous. Also there is a disclaimer reminding that this site is not an alternative to therapy or other treatments. You will receive weekly emails/texts about new posts. We will track how often and how long you log-on to the site.

Content from the website will be downloaded except if it contains identifying information. In cases where there is identifying information the content will be deleted permanently.

In <u>Group 2</u> you will not get access to log-on to the site. You will instead be asked to read a publicly available SOVA article, and then you will be asked to respond to a discussion question about what you read, using the REDCap survey website. What you write will only be viewed by the research team. You will be asked to do this once a month for three months.

In both of the groups, you will take online surveys using the REDCap website. These surveys will contain questions about demographics (like your age, education), experiences with discrimination, your feedback on whether the intervention and study are acceptable to you, and questions about self-esteem, mental health, social support, loneliness, and stigma.

All survey data we collect from you is stored on a secure online survey platform called REDCap which the University of Pittsburgh has used for many years. And the data we extract from that online survey platform will be stored on a secure University of Pittsburgh server. We may share de-identified data meaning it does not have any information that can trace the data back to you (identifiers) with other researchers in the future.

If you have more questions, you can contact us at the study email, sovalab@pitt.edu. If you have questions about your rights as a research participant, you can contact the Human Subject Protection Advocate at the University of Pittsburgh IRB (Institutional Review Board) Office at 866.212.2668.

## **RISKS**

We don't expect that there are any major risks to you for participating in this study.

There may be some minor risks, the main one being in the situation that someone obtains confidential information about you. To prevent that, we will take several steps. We use a secure survey platform called REDCap. Data we take from REDCap will be stored on Pitt secured OneDrive.

The email and mobile phone you provide will be used for communication about the study and reminding about study tasks and surveys. Text messages may not be encrypted or secure during their transmission or storage and it is possible they could be intercepted and used by others not associated with this study. We advise that you do not send identifiable information via text.

Emails may not be encrypted during transmission or storage and may be intercepted and used by others not associated with this study. We advise you to ensure to password protect your email. We also encourage you to lock and password protect your smartphone to ensure privacy.

Another risk is feeling embarrassed when answering questions during the survey. We encourage you to only answer questions you feel comfortable with.

## **BENEFITS**

While there may not be a direct benefit for participating in the research study, we will provide you with crisis resources at the end, which you might find helpful. If you have questions about anything we have discussed, we can do our best to answer them.

### **PAYMENTS**

You will receive \$25 for each survey at baseline, at 6 weeks, and at 3 months. Intervention completion

For Group 1 (SOVA Ambassador arm) you will receive \$10/month if you create content for the site at least one time a month and an additional \$5/month for comments written on the website in response to a different article.

For Group 2 you will receive \$10/month if you write at least one comment in response to a discussion question and an additional \$5/month if you answer a second discussion question.

All participants who participate in all parts of the study (\$75 total for surveys, \$45 total for intervention full participation) can receive up to \$120 for participating in all parts of the study on a pre-paid gift card.

## CONFIDENTIALITY

We do our best to keep all information on the website anonymous. Participants are counseled to not put any identifying information on the website. Anything you tell us in the survey or intervention will remain confidential. We will download text from the website and REDCap which we may analyze as research data. To protect your confidentiality, any information that might identify you, your family, friends, or others will be removed.

To help us protect your privacy, we have a Certificate of Confidentiality from the National Institutes of Health. This Certificate means Dr. Radovic and her team can legally refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

The Certificate cannot be used to resist a demand for information from personnel of the United States Government that is used for auditing or evaluation of federally-funded projects or for information that must be disclosed to meet the requirements of the federal Food and Drug Administration (FDA).

You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written assent to receive research information, then the researchers may not use the Certificate to withhold that information.

The Certificate of Confidentiality will not be used to prevent disclosure to state or local authorities of child abuse and neglect or harm to self or others.

If during the course of the research activities we believe that you are a risk to yourself or others we may contact your parent.

The data we obtain for this study may be shared with other groups such as the National Institutes of Health, UPMC Children's Hospital of Pittsburgh, and the University of Pittsburgh Office of Research Protections.

Information collected from this study may be shared with other investigators interested in this topic; however, this information will be shared in a de-identified manner (i.e., without identifiers).

Your survey data may be uploaded along with all other study data to the National Data Archive (NDA), but this will be without any identifiers.

Per University of Pittsburgh policy all research records must be maintained for at least 7 years following final reporting or publication of a project. For projects involving minors, records must be maintained until child participants reach the age of 25.

#### WITHDRAW

Participation in this research study is entirely voluntary. If at any point in the survey you don't want to answer a question, we can skip it, and if you want to stop the survey or continue it later, that is fine, too. Whether or not you participate is up to you. You may withdraw from the study at any time and there is no penalty for withdrawal.

## ASSENT TO PARTICIPATE

I understand that I am encouraged to ask questions, voice concerns or complaints about any part of this research study during this study. Any future questions, concerns or complaints will be answered by a qualified individual or by the investigator(s) listed on the first page of this assent document at the telephone number(s) given. I understand that I may always request that my questions, concerns or complaints be addressed by a listed investigator. I understand that I may contact the Human Subjects Protection Advocate of the Human Research Protection office, University of Pittsburgh (1-866-212-2668) to discuss problems, concerns, and questions; obtain information; offer input; or discuss situations that occurred during my participation. By typing my full name, date of birth, and the school I go to (or went to most recently), I assent to participate in this research study.

# CONSENT TO ACT AS A PARTICIPANT IN A RESEARCH STUDY

Do you assent to participate in the study? (yes/no)

What is the name of the school you currently or most recently attended?

What is your date of birth?

Type your full name: